CLINICAL TRIAL: NCT00117117
Title: A Study to Assess Symptom Burden in Subjects With Nonmyeloid Malignancies Receiving Chemotherapy and Aranesp®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020132
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Anemia
Keywords: Chemotherapy induced anemia; Amgen; Aranesp®; darbepoetin alfa
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp

SUMMARY:
The purpose of this trial is to prospectively assess the relationship between changes in hemoglobin (hgb) and changes in symptom burden associated with anemia in cancer patients receiving chemotherapy supported with Aranesp®.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with nonmyeloid malignancy(ies)
* Anemia (hgb less than or equal to 11.0 g/dL) due to cancer and chemotherapy

Exclusion Criteria:

* Subjects with acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML), myelodysplastic syndromes (MDS)
* Unstable cardiac disease or anemia due to other causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2423
Dates: Start 2002-09; Study Completion 2003-12

PRIMARY OUTCOMES:
Patient reported outcomes

SECONDARY OUTCOMES:
Changes in hemoglobin endpoints and RBC transfusion requirements

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Gregory SA. Efficacy of Darbepoetin Alfa in the Treatment of Chemotherapy-Induced Anemia in Non-Hodgkin's Lymphoma. Support Cancer Ther. 2006 Jul 1;3(4):232-9. doi: 10.3816/SCT.2006.n.021. PMID 18632499
- [Result] Gabrilove JL, Perez EA, Tomita DK, Rossi G, Cleeland CS. Assessing symptom burden using the M. D. Anderson symptom inventory in patients with chemotherapy-induced anemia: results of a multicenter, open-label study (SURPASS) of patients treated with darbepoetin-alpha at a dose of 200 microg every 2 weeks. Cancer. 2007 Oct 1;110(7):1629-40. doi: 10.1002/cncr.22943. PMID 17694552
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com